CLINICAL TRIAL: NCT02817568
Title: The Evaluation of MCP-1 and CCR-2 Gene Polymorphisms Frequency and The Effects of This Polymorphism on Gene Expression in Patients With Aggressive Periodontitis
Brief Title: Frequency Of MCP-1 And CCR2 Gene Polymorphisms And Its Effect On Gene Expression In Patients With AgP
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Collaborators: Selcuk University (Other)
Responsible Party: Principal Investigator, Sadiye Gunpinar, Abant Izzet Baysal University, Faculty of Dentistry, Abant Izzet Baysal University
Other Study IDs: 11102024; SU1985 (Other: SelcukUniversity); SUPeriodontology (Other: SelcukUniversity)
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Aggressive Periodontitis
Keywords: Aggressive Periodontitis; C-C chemokine receptor 2; Gene expression; monocyte chemoattractant protein-1,; restriction fragment length polymorphism
MeSH Terms: conditions — Aggressive Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral Blood of each subject is kept -80 celcius for further analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Aggressive Periodontitis (case): Single intervention has been performed for each subject. Peripheral blood sample was obtained in conjunction with clinical measurements in this intervention.(Drawing Blood)
  Interventions: Other: Drawing Blood
- Healthy (Control): Single intervention has been performed for each subject. Peripheral blood sample was obtained in conjunction with clinical measurements in this intervention. (Drawing Blood)
  Interventions: Other: Drawing Blood

INTERVENTIONS:
Other: Drawing Blood — Drawing Blood for genetic analysis

SUMMARY:
The aim of this study is to estimate genetic impact of MCP-1 -2518 and its receptor CCR2 -190 polymorphisms on AgP patients among Turkish individuals and whether MCP-1 genotype effects mRNA levels of Peripheral Blood Mononuclear Cell Leukocyte (PBML)

DETAILED DESCRIPTION:
Differences in structure of gene or non genetic factors such as nutrition/environmental factors may alter functional gene product: mRNA/protein which play crucial roles in immune system. This can lead developing defective immune responses, exacerbation of current inflammation and increased host susceptibility to inflammatory diseases. Monocyte functions can be critical with regard to getting individuals susceptible to periodontitis. Similarly Garrison and Nichols (1989) reported that hyper-inflammatory monocyte phenotype can be deterministic in periodontal destruction. For this reason, regulation of MCP-1 and CCR2 expression, which have an essential role in defense system, may be a crucial step for managing inflammatory diseases as well as periodontitis.

Because of complex genetic nature of periodontal disease, we hypothesized that gene polymorphisms of MCP-1 and CCR2 could be associated with AgP and could alter the production of functional proteins, as a result might influence the susceptibility. Therefore, the primary aim of this study was to estimate genetic impact of MCP-1 and its receptor CCR2 polymorphisms on AgP patients among Turkish individuals and secondary outcome was whether MCP-1 genotype effects mRNA levels of PBML.

A total of 215 Turkish subjects from inner Anatolia including, 108 Aggressive periodontitis (AgP) and 107 age, gender and ethnic matched periodontally healthy (H) controls were recruited in this cross-sectional case control study. The control group included periodontally healthy volunteers from staff and other subjects referring to the School of Dentistry. The diagnosis of subjects were established on the basis of clinical and radiographic examination. Periodontally H control group (n:107) had <3mm probing Depth (PD), <2 gingival Index (GI) and no signs of interproximal attachment loss and a history of periodontal disease. Patients with AgP (n:108) were diagnosed by the 1999 International World Workshop for a Classification of Periodontal Diseases and Conditions. The AgP group included individuals diagnosed with localized AgP (LAgP) or generalized AgP (GAgP) who were otherwise healthy. Periodontal attachment loss ≥4 mm not involving more than two permanent teeth, other than the first molars and incisors were diagnosed with LAgP (n: 43); patients with involvement of at least three teeth, other than the first molars and incisors with an attachment loss ≥4 mm were diagnosed with GAgP (n: 65) Genomic DNA was isolated from a peripheral blood sample obtained from each subject. Gene polymorphisms of MCP-1 -2518 A/G and CCR2 -190 G/A were analyzed by a standard polymerase chain reaction-restriction fragment length polymorphism (PCR-RFLP) assay. Gene expression levels were quantified in peripheral blood leukocytes from 25 AgP and 15 periodontally H controls by quantitative real-time PCR. Threshold cycles (Ct ) values obtained from the RT-PCR analysis based on SYBR Green detection and data was normalized via ΔC t .

Sample size was determined by power analysis prior to study. According to this; an expected difference 20% in allele frequencies with 80% power, and % 95 confidence interval it was calculated that minimum of 102 patients were necessary in each group with a significance level of 0.05. ( ⃰ G. Power: 3.1.2). When comparing the numeric characteristics between H and AgP groups,non-parametric Mann-Whitney U test; between H, LAgP and GAgP groups then Kruskal Wallis with Bonferroni correction were calculated.

Deviations from Hardy-Weinberg equilibrium were assessed in the H and AgP groups based on genotype distribution for MCP-1 -2518 and CCR2 -190 by using a chi-squared test. The differences in genotype and allele frequencies between groups were also detected by the chi-square test. We used independent samples t-test for comparison of gene expression levels between groups and one way ANOVA was used to determine the effect of MCP-1 -2518 genotype on gene expression, based on log-transformed data. Significance level was P = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Periodontally H control group had < 3mm PD, < 2 GI and no signs of interproximal attachment loss and a history of periodontal disease.
* The AgP group included individuals diagnosed with localized AgP (LAgP) or generalized AgP (GAgP) who were otherwise healthy. Periodontal attachment loss ≥4 mm not involving more than two permanent teeth, other than the first molars and incisors were diagnosed with LAgP (n: 43); patients with involvement of at least three teeth, other than the first molars and incisors with an attachment loss ≥4 mm were diagnosed with GAgP

Exclusion Criteria:

* Patients who have any systemic diseases or conditions that could effect the periodontium
* hepatitis and/or immunodeficiency virus infection
* a history of periodontal treatment and antibiotic therapy within the 6 months
* < 16 teeth in their mouth
* Subjects who had smoked and were ongoing orthodontic treatment were excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This cross-sectional case control study was carried out at Selcuk University, Faculty of Dentistry, Department of Periodontology. The control group included periodontally healthy volunteers from staff and other subjects referring to the School of Dentistry.
Sampling Method: Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Frequency of MCP-1 -2518 A/G and CCR2 -190 G/A gene polymorphisms in Aggressive Periodontitis | one year

SECONDARY OUTCOMES:
MCP-1 gene expression in AgP patients | six months

CONTACTS AND LOCATIONS:
Overall Officials: Nilgun O Alptekin, Phd, DDS, Principal Investigator — Baskent University, Faculty of Dentistry, Periodontology Department; Sadiye Gunpinar, Phd, DDS, Principal Investigator — Abant Izzet Baysal University, Faculty of Dentistry, Periodontology Department; Hasan Acar, Phd, Principal Investigator — Selcuk University, Faculty of Medicine, Department of Genetics; Vasfiye B Ucar, Phd, Principal Investigator — Selcuk University, Faculty of Medicine, Department of Genetics

IPD SHARING:
Plan to Share IPD: No
Individual participant data is kept in private computer and all data can be shared if necessary

REFERENCES:
- [Background] Armitage GC. Periodontal diagnoses and classification of periodontal diseases. Periodontol 2000. 2004;34:9-21. doi: 10.1046/j.0906-6713.2002.003421.x. No abstract available. PMID 14717852
- [Result] Yu X, Graves DT. Fibroblasts, mononuclear phagocytes, and endothelial cells express monocyte chemoattractant protein-1 (MCP-1) in inflamed human gingiva. J Periodontol. 1995 Jan;66(1):80-8. doi: 10.1902/jop.1995.66.1.80. PMID 7891256
- [Result] Zhu XL, Meng HX, Zhang L, Xu L, Chen ZB, Shi D, Feng XH, Zhang X. Association analysis between the -2518MCP-1(A/G) polymorphism and generalized aggressive periodontitis in a Chinese population. J Periodontal Res. 2012 Jun;47(3):286-92. doi: 10.1111/j.1600-0765.2011.01426.x. Epub 2011 Nov 27. PMID 22117820
- [Result] Pradeep AR, Daisy H, Hadge P. Gingival crevicular fluid levels of monocyte chemoattractant protein-1 in periodontal health and disease. Arch Oral Biol. 2009 May;54(5):503-9. doi: 10.1016/j.archoralbio.2009.02.007. Epub 2009 Mar 16. PMID 19286166
- [Result] Emingil G, Atilla G, Huseyinov A. Gingival crevicular fluid monocyte chemoattractant protein-1 and RANTES levels in patients with generalized aggressive periodontitis. J Clin Periodontol. 2004 Oct;31(10):829-34. doi: 10.1111/j.1600-051X.2004.00584.x. PMID 15367184
- [Result] Kurtis B, Tuter G, Serdar M, Akdemir P, Uygur C, Firatli E, Bal B. Gingival crevicular fluid levels of monocyte chemoattractant protein-1 and tumor necrosis factor-alpha in patients with chronic and aggressive periodontitis. J Periodontol. 2005 Nov;76(11):1849-55. doi: 10.1902/jop.2005.76.11.1849. PMID 16274303